CLINICAL TRIAL: NCT01839422
Title: Functionnal Magnetic Resonnance Imaging (fMRI)Study of Cerebral Substrates of New Musical and Pictorial Learning in Alzheimer Patients
Brief Title: Imaging of New Learning in Severe Alzheimer's Disease Patients
Acronym: INCAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-A00351-40
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Controls (Experimental): Memory assessment. Brain imaging examination MRI.
  Interventions: Behavioral: Memory assessment; Other: Brain imaging examination MRI
- Beginner Alzheimer's Disease patients (Experimental): Memory assessment. Brain imaging examination MRI.
  Interventions: Behavioral: Memory assessment; Other: Brain imaging examination MRI
- Severe Alzheimer's Disease patients (Experimental): Memory assessment. Brain imaging examination MRI.
  Interventions: Behavioral: Memory assessment; Other: Brain imaging examination MRI

INTERVENTIONS:
Behavioral: Memory assessment — Cognitive assessment : Neuropsycological tests, learning sessions of new stimuli.
Other: Brain imaging examination MRI — Brain imaging examination : Structural and functional MRI to compare differences between each sample.

SUMMARY:
This research attempts to better understand the altered and preserved memory mechanisms in Alzheimer disease, particularly to better apprehend learning implicit memory processes, and give a scientific support to non-pharmalogical interventions. At the present time, it is possible to delay the emergence of the symptoms related to this disease, eventually to decrease it, but not to cure it. Yet, care these patients became a crucial question and the solutions proposed to healthy aging people are not appropriate for Alzheimer patients who present specific disorders. The improvement of the quality of life of the institutionalized patients lies on a better comprehension of their disorders but also of their preserved abilities. The literature testifies of a great heterogeneity in the clinical expression of this disease, however we noticed two constants with regard to the capabilities generally announced as being preserved, on one hand, the implicit memory, and on the other hand the artistic aptitudes, and more particularly musical capabilities.

Patients with Alzheimer disease present a particularly severe and early deterioration of episodic memory. Thus, at the beginning of the disease the explicit acquisition of new knowledge becomes increasingly difficult. However, some clinical observations, such as new learning of unknown songs, even with patients at a severe stage of the illness, seem to support the assumption of a preservation of some implicit learning abilities. Indeed, several studies already showed preserved implicit memory capabilities among patients with Alzheimer disease, mostly at the beginning stage of the illness: preserved effects of perceptual priming, procedural learning. Thus, we are mainly interested by the effects of exposure and the rising of a feeling of familiarity, both showing preserved implicit learning abilities, for moderate to severe Alzheimer patients. However, no study was carried out to date using the neuroimaging techniques, among Alzheimer patients at a moderated to severe stage of illness, with the main objective to identify the cerebral substrates implied in the learning of new knowledge.

Indeed, several studies already showed preserved implicit memory capabilities among patients with Alzheimer disease, mostly were performed at the beginning stage of the illness and none of them have studied theses learning abilities for moderate to severe Alzheimer patients.

The objective of this work is to specify, in severe form of Alzheimer disease, the cognitive mechanisms allowing the memorizing (feeling of familiarity) of new information and thus to highlight neural networks underlying this learning process (recently learned stimuli vs old stimuli). The goal is to propose a positive image of the Alzheimer patients, in understanding which cognitive mechanisms and cerebral areas allow these learning capabilities.

20 patients Alzheimer at a moderate to severe stage, 20 patients at a mild to moderate stage of the illness, and 20 healthy aging participants, are selected after a neurological interview and a neuropsychological evaluation. The whole of the included participants take part of the experimental protocol organized in two phases: - the phase of familiarization and the phase of test. The phase of familiarization consists of the repeated exposure (daily session before the MRI acquisition) of new songs and new painting until obtaining a high feeling of familiarity for each item. The phase of test is carried out in the 3T MRI camera, it comprises an anatomical (T1, T2 MRI) and a functional acquisitions. The functional acquisition corresponds to a passive listening and seeing tasks of musical and pictorial stimuli. Finally, all participants realize a debriefing phase that allows obtaining a feedback on the familiarity of stimuli presented during the functional acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Native language: French
* Medical, neurological, neuropsychological and neuroradiological depth in accordance with the criteria for inclusion and exclusion-specific population, that is to say:

  * Healthy Elderly volunteers: over 60 years old, living at home, without memory complaints, normal performances compared to the age and the educational level for all tests of the diagnostic battery.
  * Alzheimer's patients: presenting the standard criteria of NINCDS-ADRDA probable Alzheimer's disease, including abnormal global cognitive function and deficits in at least two cognitive domains identified by the diagnostic battery.

Exclusion Criteria:

* The sudden onset of cognitive impairments (as opposed to their slow and gradual installation in Alzheimer's disease)
* A chronic neurological, psychiatric, endocrine, hepatic or infectious complaint
* A history of major disease (an uncontrolled diabetes, a lung, heart, metabolic, hematologic, endocrine disease or a severe cancer);
* A medication that may interfere with memory or metabolic measures
* A alcohol or drugs abuse
* The cons-indications to MRI (claustrophobia, metallic object in the body).
* A predominantly left-hand (score below 50% in Edinburgh Inventory)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Succesful learning of new songs and paintings, succesful MRI acquisitions. | 10 days max. One week for the learning sessions, before MRI scans done one or two days after.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent de La Sayette, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- GIP Cyceron, Caen, France